CLINICAL TRIAL: NCT05843058
Title: The Effect of Laughter Yoga on Psychological Wellness on Women With Gynecological Cancer
Brief Title: The Effect of Laughter Yoga on Psychological Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, kerime derya beydağ, Assoc. Prof., Istanbul Gedik University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DBEYDAG002*
Record Dates: First submitted 2023-03-30; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Laughter; Gynecologic Cancer; Psychological
MeSH Terms: conditions — Laughter | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laughter yoga (Experimental): The psychological well-being scale was filled in at the first encounter with the patient. Then, 12 sessions of laughter yoga were performed and after 12 sessions, the psychological well-being scale was applied again.(Laughter yoga was practiced twice a week for 6 weeks)
  Interventions: Behavioral: laughter yoga
- Standard care (No Intervention): The psychological well-being scale was filled in at the first encounter with the patient. Then, 6 weeks later, the psychological well-being scale was applied again.

INTERVENTIONS:
Behavioral: laughter yoga — The effect of laughter yoga on psychologıcal wellness ın women wıth gynecologıcal cancer has been evaluated.
  Arms: laughter yoga

SUMMARY:
The aim of the thesis is to determine the effect of laughter yoga on psychological well-being in women diagnosed with Gynecological Cancer.The population of the study consists of the patients registered in the oncology service of Tepecik Training and Research Hospital in Izmir. The study was carried out with 70 patients, 35 of which were interventions and 35 controls, who were treated in the oncology service of Izmir Tepecik Training and Research Hospital.

DETAILED DESCRIPTION:
The aim of the thesis is to determine the effect of laughter yoga on psychological well-being in women diagnosed with Gynecological Cancer.The population of the study consists of the patients registered in the oncology service of Tepecik Training and Research Hospital in Izmir. The study was carried out with 70 patients, 35 of which were interventions and 35 controls, who were treated in the oncology service of Izmir Tepecik Training and Research Hospital between October 1, 2021 and April 1, 2022. In order to measure the effect of laughter yoga on psychological well-being, the Psychological Well-Being Scale was applied to both the experimental group and the control group patients.

ELIGIBILITY:
Inclusion Criteria:

* • Volunteering to participate in the study

  * Having the ability to read, write, speak and understand Turkish
  * Being diagnosed with gynecological cancer
  * Being in Stage II or Stage III of the gynecological cancer staging processes
  * The patient's internet access

Exclusion Criteria:

* The patient is Stage 4
* Lack of internet access

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — WOMEN WITH GYNECOLOGICAL CANCER
Enrollment: 70 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Psychological well-being scale (PWS) | 6 months
  Change in Psychological well-being scale (PWS); is a 7-point Likert type scale ranging from strongly disagree (1) to strongly agree (7). All items are expressed positively. The lowest score is 8 and the highest score is 56. A high score indicates that the individual has many psychological resources and strengths.
  The effect of laughter yoga on psychologıcal wellness.

CONTACTS AND LOCATIONS:
Overall Officials: Kerime Derya BEYDAG, Study Director — https://akademik.yok.gov.tr/AkademikArama/view/viewAuthor.jsp
Locations (1):
- Kerime Derya BEYDAG, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bennett PN, Hussein WF, Reiterman M, Yu J, Schiller B. The effects of laughter therapy on depression symptoms in patients undergoing center hemodialysis: A pragmatic randomized controlled trial. Hemodial Int. 2020 Oct;24(4):541-549. doi: 10.1111/hdi.12870. Epub 2020 Aug 25. PMID 32844575
- [Background] Cho EA, Oh HE. [Effects of laughter therapy on depression, quality of life, resilience and immune responses in breast cancer survivors]. J Korean Acad Nurs. 2011 Jun;41(3):285-93. doi: 10.4040/jkan.2011.41.3.285. Korean. PMID 21804337
- [Background] Demir Dogan M. The Effect of Laughter Therapy on Anxiety: A Meta-analysis. Holist Nurs Pract. 2020 Jan/Feb;34(1):35-39. doi: 10.1097/HNP.0000000000000363. PMID 31725098
- [Background] Ghodsbin F, Sharif Ahmadi Z, Jahanbin I, Sharif F. The effects of laughter therapy on general health of elderly people referring to jahandidegan community center in shiraz, iran, 2014: a randomized controlled trial. Int J Community Based Nurs Midwifery. 2015 Jan;3(1):31-8. PMID 25553332
- [Background] Hatzipapas I, Visser MJ, Janse van Rensburg E. Laughter therapy as an intervention to promote psychological well-being of volunteer community care workers working with HIV-affected families. SAHARA J. 2017 Dec;14(1):202-212. doi: 10.1080/17290376.2017.1402696. PMID 29169302
- [Background] Kim SH, Kim YH, Kim HJ. Laughter and Stress Relief in Cancer Patients: A Pilot Study. Evid Based Complement Alternat Med. 2015;2015:864739. doi: 10.1155/2015/864739. Epub 2015 May 24. PMID 26064177